CLINICAL TRIAL: NCT00882128
Title: Evaluation of the Control Level (GINA) of Asthmatic Patients Consulting Their General Practitioner for a Seasonal Increase of Respiratory Symptoms (High and / or Low), Whether an Inhaled Corticotherapy is Taken or Not
Brief Title: Evaluation of the Control Level of Asthmatic Patients With Seasonal Increase of Respiratory Symptoms (High and/or Low)
Acronym: SAISON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-RFR-DUM-2008/2
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Asthma; Respiratory Symptoms
Keywords: Asthma seasonal respiratory symptoms; Asthmatic patients with increase of respiratory symptoms
MeSH Terms: conditions — Asthma; Signs and Symptoms, Respiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
To evaluate the level of control of Asthma (GINA : controlled, partially controlled, not controlled) of asthmatic patients consulting their general practitioner for a seasonal increase of respiratory symptoms (high and / or low) whether an inhaled corticotherapy is taken or not.

ELIGIBILITY:
Inclusion Criteria:

* Asthmatic adults consulting for a seasonal increase of respiratory symptoms (high/low) and treated with PRN fast acting bronchodilator alone or associated with inhaled IGCS, excluding all other treatments for asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first 3 consecutive adult and asthmatic patients consulting their general practitioner for a seasonal increase of respiratory symptoms (high and / or low) and treated with PRN fast acting bronchodilatator alone or associated with inhaled IGCS, excluding all other treatments for asthma.
Sampling Method: Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2009-05; Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the control level of Asthma of asthmatic patients consulting their GP for a seasonal increase of respiratory symptoms (high/low) with an inhaled corticotherapy or not. | One shot (patients will only have one visit to attend - this visit will take place between May 09 and September 09)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Castaigne Castaigne, Study Director — AstraZeneca
Locations (1051):
- France (1051):
  - Research Site, Abbaretz
  - Research Site, Acheux-en-Amiénois
  - Research Site, Agen
  - Research Site, Agneaux
  - Research Site, Agon-Coutainville
  - Research Site, Aignay-le-Duc
  - Research Site, Aiguillon
  - Research Site, Aiserey
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Ajaccio
  - Research Site, Albi
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Alleins
  - Research Site, Allonnes
  - Research Site, Althen-des-Paluds
  - Research Site, Amagne
  - Research Site, Ambert
  - Research Site, Ambès
  - Research Site, Andance
  - Research Site, Andard
  - Research Site, Anizy-le-Château
  - Research Site, Annay
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Anzin
  - Research Site, Arc-et-Senans
  - Research Site, Arcachon
  - Research Site, Arches
  - Research Site, Argentat
  - Research Site, Argenteuil
  - Research Site, Arles
  - Research Site, Art-sur-Meurthe
  - Research Site, Arthez-de-Béarn
  - Research Site, Asnières-sur-Seine
  - Research Site, Aspiran
  - Research Site, Aubagne
  - Research Site, Aubervilliers
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Auchy-les-Mines
  - Research Site, Audincourt
  - Research Site, Augny
  - Research Site, Aulnat
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aumetz
  - Research Site, Aurillac
  - Research Site, Auterive
  - Research Site, Authon-du-Perche
  - Research Site, Autun
  - Research Site, Auxerre
  - Research Site, Auxi-le-Château
  - Research Site, Auxonne
  - Research Site, Auzon
  - Research Site, Avallon
  - Research Site, Avignon
  - Research Site, Avoine
  - Research Site, Axat
  - Research Site, Bachant
  - Research Site, Badevel
  - Research Site, Bagneux
  - Research Site, Baignes Ste Radegonde
  - Research Site, Baigneux-les-Juifs
  - Research Site, Bailly-Romainvilliers
  - Research Site, Bains
  - Research Site, Bais
  - Research Site, Balan
  - Research Site, Bannalec
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Barentin
  - Research Site, Basse-Goulaine
  - Research Site, Bassens
  - Research Site, Baulon
  - Research Site, Bayeux
  - Research Site, Bayonne
  - Research Site, Beaucaire
  - Research Site, Beauchamp
  - Research Site, Beaumesnil
  - Research Site, Beaumont-de-Pertuis
  - Research Site, Beaumont-en-Véron
  - Research Site, Beaumont-sur-Lèze
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Beauvallon
  - Research Site, Beauzelle
  - Research Site, Behren-lès-Forbach
  - Research Site, Belfort
  - Research Site, Bellemene
  - Research Site, Belleville-sur-Meuse
  - Research Site, Bellême
  - Research Site, Belz
  - Research Site, Benquet
  - Research Site, Berck
  - Research Site, Bergbieten
  - Research Site, Bergholtz
  - Research Site, Bermerain
  - Research Site, Berson
  - Research Site, Besançon
  - Research Site, Bethoncourt
  - Research Site, Bezons
  - Research Site, Bérat
  - Research Site, Bétaille
  - Research Site, Béthisy-Saint-Pierre
  - Research Site, Béville-le-Comte
  - Research Site, Béziers
  - Research Site, Biganos
  - Research Site, Billom
  - Research Site, Biver
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanquefort
  - Research Site, Blénod-lès-Pont-à-Mousson
  - Research Site, Bobigny
  - Research Site, Boëge
  - Research Site, Boën-sur-Lignon
  - Research Site, Bois-en-Ardres
  - Research Site, Bois-le-Roi
  - Research Site, Bolbec
  - Research Site, Bollène
  - Research Site, Bondoufle
  - Research Site, Bonnelles
  - Research Site, Bonnières-sur-Seine
  - Research Site, Boos
  - Research Site, Bordeaux
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bort-les-Orgues
  - Research Site, Bouffémont
  - Research Site, Bouguenais
  - Research Site, Boujan-sur-Libron
  - Research Site, Boulogne-Billancourt
  - Research Site, Boulogne-sur-Gesse
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourcefranc-le-Chapus
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourges
  - Research Site, Bourron-Marlotte
  - Research Site, Bourth
  - Research Site, Boves
  - Research Site, Boynes
  - Research Site, Branne
  - Research Site, Brantôme
  - Research Site, Bresles
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Bretteville-l'Orgueilleuse
  - Research Site, Bréhal
  - Research Site, Briançon
  - Research Site, Brie-Comte-Robert
  - Research Site, Brignais
  - Research Site, Brignoles
  - Research Site, Brive-la-Gaillarde
  - Research Site, Brunstatt
  - Research Site, Bruyères-sur-Oise
  - Research Site, Buc
  - Research Site, Bulgnéville
  - Research Site, Bussang
  - Research Site, Cachan
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cahuzac-sur-Vère
  - Research Site, Calais
  - Research Site, Calvi
  - Research Site, Calvisson
  - Research Site, Camblanes
  - Research Site, Cambrai
  - Research Site, Camors
  - Research Site, Canteleu
  - Research Site, Cany-Barville
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Cappelle-en-Pévèle
  - Research Site, Cappelle-la-Grande
  - Research Site, Carantec
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carhaix-Plouguer
  - Research Site, Carpentras
  - Research Site, Carquefou
  - Research Site, Carresse-Cassaber
  - Research Site, Carvin
  - Research Site, Castelnau-Montratier
  - Research Site, Castets-en-Dorthe
  - Research Site, Caveirac
  - Research Site, Caylus
  - Research Site, Celles-sur-Plaine
  - Research Site, Cérences
  - Research Site, Cérilly
  - Research Site, Chabris
  - Research Site, Chaingy
  - Research Site, Chalais
  - Research Site, Chalamont
  - Research Site, Chaleins
  - Research Site, Chambéry
  - Research Site, Champagne-sur-Oise
  - Research Site, Champagne-sur-Seine
  - Research Site, Champagnole
  - Research Site, Champcueil
  - Research Site, Champdeniers-Saint-Denis
  - Research Site, Champeaux
  - Research Site, Champigneulles
  - Research Site, Champigné
  - Research Site, Champigny-sur-Marne
  - Research Site, Champs-sur-Marne
  - Research Site, Chanteheux
  - Research Site, Chantepie
  - Research Site, Chantilly
  - Research Site, Chantonnay
  - Research Site, Chapelle Saint Martin Plaine
  - Research Site, Charleville-Mézières
  - Research Site, Charmes
  - Research Site, Chartres
  - Research Site, Chasseneuil-du-Poitou
  - Research Site, Chassieu
  - Research Site, Chateauneuf Ille Vilaine
  - Research Site, Chatte
  - Research Site, Chauvigny
  - Research Site, Châlons-en-Champagne
  - Research Site, Château-d'Olonne
  - Research Site, Châteaubriant
  - Research Site, Châteaugay
  - Research Site, Châteauneuf-sur-Cher
  - Research Site, Châteauroux
  - Research Site, Châtelaillon-Plage
  - Research Site, Châtellerault
  - Research Site, Châtenay-Malabry
  - Research Site, Châtenois-les-Forges
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Cherbourg Octeville
  - Research Site, Cherisy
  - Research Site, Cherves-Richemont
  - Research Site, Cheval-Blanc
  - Research Site, Chinon
  - Research Site, Choisey
  - Research Site, Cholet
  - Research Site, Ciboure
  - Research Site, Ciry-le-Noble
  - Research Site, Clairac
  - Research Site, Clamart
  - Research Site, Clermont
  - Research Site, Clermont-Ferrand
  - Research Site, Clichy
  - Research Site, Colomars
  - Research Site, Colombes
  - Research Site, Colombey-les-Belles
  - Research Site, Colomiers
  - Research Site, Combrit
  - Research Site, Combs-la-Ville
  - Research Site, Comines
  - Research Site, Commentry
  - Research Site, Communay
  - Research Site, Comps
  - Research Site, Conflans Ste Honorine
  - Research Site, Contes
  - Research Site, Conty
  - Research Site, Corbehem
  - Research Site, Corbeil-Essonnes
  - Research Site, Corbie
  - Research Site, Corcieux
  - Research Site, Cordes-sur-Ciel
  - Research Site, Coudekerque-Branche
  - Research Site, Coudes
  - Research Site, Courbevoie
  - Research Site, Courcy
  - Research Site, Courçon
  - Research Site, Courpière
  - Research Site, Coursan
  - Research Site, Courseulles-sur-Mer
  - Research Site, Courthézon
  - Research Site, Cousolre
  - Research Site, Coussac-Bonneval
  - Research Site, Coutances
  - Research Site, Coutouvre
  - Research Site, Coye-la-Forêt
  - Research Site, Cravanche
  - Research Site, Creil
  - Research Site, Creysse
  - Research Site, Crécy-la-Chapelle
  - Research Site, Créteil
  - Research Site, Croissy-sur-Seine
  - Research Site, Croix
  - Research Site, Crolles
  - Research Site, Crosne
  - Research Site, Cuers
  - Research Site, Cugand
  - Research Site, Cuise-la-Motte
  - Research Site, Dambach-la-Ville
  - Research Site, Daoulas
  - Research Site, Daux
  - Research Site, Décines-Charpieu
  - Research Site, Dieppe
  - Research Site, Dieuze
  - Research Site, Digne-les-Bains
  - Research Site, Dinard
  - Research Site, Dissay
  - Research Site, Dole
  - Research Site, Dompierre-sur-Mer
  - Research Site, Donges
  - Research Site, Dossenheim-sur-Zinsel
  - Research Site, Dugny-sur-Meuse
  - Research Site, Dunières
  - Research Site, Dunkirk
  - Research Site, Eaubonne
  - Research Site, Ennezat
  - Research Site, Entre Deux
  - Research Site, Envermeu
  - Research Site, Eragny Sur Oise
  - Research Site, Escaudain
  - Research Site, Esquerdes
  - Research Site, Estivareilles
  - Research Site, Eygalières
  - Research Site, Eyguières
  - Research Site, Échirolles
  - Research Site, Écuisses
  - Research Site, Épernay
  - Research Site, Épieds-en-Beauce
  - Research Site, Épierre
  - Research Site, Épinal
  - Research Site, Épinay-sur-Seine
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étalondes
  - Research Site, Évin-Malmaison
  - Research Site, Évreux
  - Research Site, Ézy-sur-Eure
  - Research Site, Fabrezan
  - Research Site, Falaise
  - Research Site, Fameck
  - Research Site, Félines
  - Research Site, Figeac
  - Research Site, Fillinges
  - Research Site, Firmi
  - Research Site, Firminy
  - Research Site, Fitilieu
  - Research Site, Flers
  - Research Site, Fléville-devant-Nancy
  - Research Site, Flize
  - Research Site, Florange
  - Research Site, Florensac
  - Research Site, Folembray
  - Research Site, Fonbeauzard
  - Research Site, Fonsorbes
  - Research Site, Fontaine
  - Research Site, Fontaine-Notre-Dame
  - Research Site, Fontenilles
  - Research Site, Fos-sur-Mer
  - Research Site, Fourneaux
  - Research Site, Foussais-Payré
  - Research Site, Francheville
  - Research Site, Franconville
  - Research Site, Fréjus
  - Research Site, Fromentine
  - Research Site, Frotey-lès-Vesoul
  - Research Site, Fumay
  - Research Site, Gaillefontaine
  - Research Site, Gaillon
  - Research Site, Gallardon
  - Research Site, Ganges
  - Research Site, Gannat
  - Research Site, Gauriac
  - Research Site, Gelles
  - Research Site, Geneuille
  - Research Site, Gennevilliers
  - Research Site, Gémenos
  - Research Site, Gémozac
  - Research Site, Générac
  - Research Site, Gif-sur-Yvette
  - Research Site, Gimont
  - Research Site, Gironde-sur-Dropt
  - Research Site, Givors
  - Research Site, Gonfaron
  - Research Site, Gonfreville-lOrcher
  - Research Site, Goudelin
  - Research Site, Gournay-en-Bray
  - Research Site, Gramat
  - Research Site, Grandcamp-Maisy
  - Research Site, Grande-Synthe
  - Research Site, Grane
  - Research Site, Gratentour
  - Research Site, Graulhet
  - Research Site, Grenoble
  - Research Site, Gréasque
  - Research Site, Gréoux-les-Bains
  - Research Site, Grièges
  - Research Site, Grignols
  - Research Site, Grimaud
  - Research Site, Guarbecque
  - Research Site, Guenrouet
  - Research Site, Guerlesquin
  - Research Site, Guérande
  - Research Site, Guéret
  - Research Site, Guidel
  - Research Site, Guise
  - Research Site, Gujan-Mestras
  - Research Site, Gy
  - Research Site, Hardelot-Plage
  - Research Site, Harnes
  - Research Site, Hazebrouck
  - Research Site, Herblay-sur-Seine
  - Research Site, Hermonville
  - Research Site, Hombourg-Haut
  - Research Site, Horbourg-Wihr
  - Research Site, Houilles
  - Research Site, Houplines
  - Research Site, Hulluch
  - Research Site, Husseren-Wesserling
  - Research Site, Hyères
  - Research Site, Igé
  - Research Site, Igoville
  - Research Site, Illiers-Combray
  - Research Site, Is-sur-Tille
  - Research Site, Isle
  - Research Site, Issoire
  - Research Site, Issoudun
  - Research Site, Issy-les-Moulineaux
  - Research Site, Ivry-sur-Seine
  - Research Site, Jacou
  - Research Site, Jeumont
  - Research Site, Joinville-le-Pont
  - Research Site, Jouars-Pontchartrain
  - Research Site, Joué-lès-Tours
  - Research Site, Jouy-le-Châtel
  - Research Site, Juniville
  - Research Site, Jurançon
  - Research Site, Jussey
  - Research Site, Juvigné
  - Research Site, Knutange
  - Research Site, L'Ardoise
  - Research Site, L'Escarène
  - Research Site, L'Haÿ-les-Roses
  - Research Site, L'Isle-d'Abeau
  - Research Site, L'Île-Saint-Denis
  - Research Site, La Bâtie-Neuve
  - Research Site, La Bouilladisse
  - Research Site, La Bretagne
  - Research Site, La Chapelle-des-Marais
  - Research Site, La Courneuve
  - Research Site, La Ferté-Saint-Aubin
  - Research Site, La Forêt-sur-Sèvre
  - Research Site, La Garde
  - Research Site, La Garenne-Colombes
  - Research Site, La Garnache
  - Research Site, La Gaude
  - Research Site, La Grande-Motte
  - Research Site, La Haye-Pesnel
  - Research Site, La Jubaudière
  - Research Site, La Loupe
  - Research Site, La Madeleine
  - Research Site, La Mézière
  - Research Site, La Motte-Servolex
  - Research Site, La Mure
  - Research Site, La Possession
  - Research Site, La Réole
  - Research Site, La Roche-en-Brenil
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Teste-de-Buch
  - Research Site, La Trinité-sur-Mer
  - Research Site, La Vraie-Croix
  - Research Site, La Walck
  - Research Site, Labastide-Murat
  - Research Site, Labenne
  - Research Site, Lacrouzette
  - Research Site, Lagarde-Enval
  - Research Site, Lagnieu
  - Research Site, Laissac
  - Research Site, Lamballe
  - Research Site, Lambersart
  - Research Site, Lambres
  - Research Site, Landerneau
  - Research Site, Landéan
  - Research Site, Landivisiau
  - Research Site, Landouge
  - Research Site, Landrecies
  - Research Site, Langeac
  - Research Site, Lanildut
  - Research Site, Lanmeur
  - Research Site, Lanouaille
  - Research Site, Lapugnoy
  - Research Site, Laroquebrou
  - Research Site, Lasseube
  - Research Site, Lathus-Saint-Rémy
  - Research Site, Latresne
  - Research Site, Lattes
  - Research Site, Laval
  - Research Site, Lavelanet
  - Research Site, Le Bouscat
  - Research Site, Le Breuil-en-Auge
  - Research Site, Le Cannet
  - Research Site, Le Cheylard
  - Research Site, Le Clion-sur-Mer
  - Research Site, Le Grand-Lemps
  - Research Site, Le Grand-Lucé
  - Research Site, Le Guillaume
  - Research Site, Le Havre
  - Research Site, Le Lardin-Saint-Lazare
  - Research Site, Le Lavandou
  - Research Site, Le Lion-dAngers
  - Research Site, Le Mans
  - Research Site, Le Mont-Dore
  - Research Site, Le Perray-en-Yvelines
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Petit Clamart
  - Research Site, Le Piton Saint Leu
  - Research Site, Le Port
  - Research Site, Le Pradet
  - Research Site, Le Raincy
  - Research Site, Le Relecq-Kerhuon
  - Research Site, Le Rouret
  - Research Site, Le Russey
  - Research Site, Le Trait
  - Research Site, Le Veurdre
  - Research Site, Lembach
  - Research Site, Lens
  - Research Site, Les Forges
  - Research Site, Les Lilas
  - Research Site, Les Lucs-sur-Boulogne
  - Research Site, Les Martres-de-Veyre
  - Research Site, Les Mées
  - Research Site, Les Mureaux
  - Research Site, Les Pieux
  - Research Site, Les Pujols
  - Research Site, Lesquin
  - Research Site, Levallois-Perret
  - Research Site, Lédignan
  - Research Site, Lézardrieux
  - Research Site, Libourne
  - Research Site, Lieu Dit Carnon Plage
  - Research Site, Liévin
  - Research Site, Lignan-sur-Orb
  - Research Site, Ligny-en-Barrois
  - Research Site, Ligueil
  - Research Site, Limeray
  - Research Site, Limoux
  - Research Site, Linas
  - Research Site, Lisieux
  - Research Site, Locmiquélic
  - Research Site, Lognes
  - Research Site, Longages
  - Research Site, Longueau
  - Research Site, Lorient
  - Research Site, Lorrez-le-Bocage-Préaux
  - Research Site, Loudes
  - Research Site, Lourdes
  - Research Site, Louverné
  - Research Site, Louvigné-du-Désert
  - Research Site, Lucé
  - Research Site, Luçon
  - Research Site, Lumbres
  - Research Site, Lumes
  - Research Site, Lunel
  - Research Site, Luneray
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Lyon
  - Research Site, L’Isle-sur-le-Doubs
  - Research Site, Madonne-et-Lamerey
  - Research Site, Magland
  - Research Site, Magnac-Bourg
  - Research Site, Maignelay-Montigny
  - Research Site, Mailly-Maillet
  - Research Site, Maintenon
  - Research Site, Maisons-Alfort
  - Research Site, Maisons-Laffitte
  - Research Site, Malemort-du-Comtat
  - Research Site, Malesherbes
  - Research Site, Malo-les-Bains
  - Research Site, Mandelieu-la-Napoule
  - Research Site, Mandeure
  - Research Site, Manosque
  - Research Site, Mantes-la-Jolie
  - Research Site, Mantes-la-Ville
  - Research Site, Marciac
  - Research Site, Marcilly-en-Villette
  - Research Site, Marcq-en-Barœul
  - Research Site, Marignane
  - Research Site, Marigny
  - Research Site, Marle
  - Research Site, Marles-les-Mines
  - Research Site, Marly
  - Research Site, Marmande
  - Research Site, Marnay
  - Research Site, Marquillies
  - Research Site, Marquion
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseille
  - Research Site, Marspich
  - Research Site, Martin-Église
  - Research Site, Marvejols
  - Research Site, Mas-Grenier
  - Research Site, Massy
  - Research Site, Maubeuge
  - Research Site, Mauguio
  - Research Site, Mauléon-Licharre
  - Research Site, Mauvezin
  - Research Site, Mauzé-sur-le-Mignon
  - Research Site, Mayenne
  - Research Site, Meaux
  - Research Site, Mennecy
  - Research Site, Mennevret
  - Research Site, Mens
  - Research Site, Mensignac
  - Research Site, Merkwiller-Pechelbronn
  - Research Site, Mers-les-Bains
  - Research Site, Mertzwiller
  - Research Site, Metz
  - Research Site, Meulan-en-Yvelines
  - Research Site, Meusnes
  - Research Site, Meximieux
  - Research Site, Meylan
  - Research Site, Meyssac
  - Research Site, Mérignac
  - Research Site, Méru
  - Research Site, Mézilles
  - Research Site, Milhaud
  - Research Site, Mimizan
  - Research Site, Miribel
  - Research Site, Moissac
  - Research Site, Moissy-Cramayel
  - Research Site, Mondelange
  - Research Site, Monistrol-sur-Loire
  - Research Site, Mont-de-Marsan
  - Research Site, Mont-Saint-Martin
  - Research Site, Mont-sous-Vaudrey
  - Research Site, Montauban
  - Research Site, Montbazin
  - Research Site, Montcy-Notre-Dame
  - Research Site, Montdidier
  - Research Site, Montendre
  - Research Site, Montesson
  - Research Site, Monteux
  - Research Site, Montélimar
  - Research Site, Montfavet
  - Research Site, Montfort-en-Chalosse
  - Research Site, Montfrin
  - Research Site, Montigny-le-Bretonneux
  - Research Site, Montigny-sur-Loing
  - Research Site, Montmorency
  - Research Site, Montmorillon
  - Research Site, Montoire-sur-le-Loir
  - Research Site, Montolieu
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montrevel-en-Bresse
  - Research Site, Morhange
  - Research Site, Mouchin
  - Research Site, Mourmelon-le-Petit
  - Research Site, Moussy-le-Neuf
  - Research Site, Moutiers-les-Mauxfaits
  - Research Site, Moyaux
  - Research Site, Mugron
  - Research Site, Mulhouse
  - Research Site, Mundolsheim
  - Research Site, Mussidan
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nanteuil-en-Vallée
  - Research Site, Narbonne
  - Research Site, Neauphle-le-Château
  - Research Site, Neufchef
  - Research Site, Neuilly-lès-Dijon
  - Research Site, Neuville-en-Ferrain
  - Research Site, Neuville-lès-Dieppe
  - Research Site, Nexon
  - Research Site, Néré
  - Research Site, Nice
  - Research Site, Niederschaeffolsheim
  - Research Site, Nieul
  - Research Site, Niort
  - Research Site, Nîmes
  - Research Site, Nogent-le-Rotrou
  - Research Site, Nogent-sur-Marne
  - Research Site, Noisy-le-Grand
  - Research Site, Noisy-le-Sec
  - Research Site, Nortkerque
  - Research Site, Notre-Dame-de-Gravenchon
  - Research Site, Notre-Dame-de-Monts
  - Research Site, Notre-Dame-du-Touchet
  - Research Site, Nouan-le-Fuzelier
  - Research Site, Novalaise
  - Research Site, Noyal-sur-Vilaine
  - Research Site, Noyon
  - Research Site, Nuisement-sur-Coole
  - Research Site, Ohlungen
  - Research Site, Oignies
  - Research Site, Oissel-sur-Seine
  - Research Site, Olby
  - Research Site, Olivet
  - Research Site, Ondres
  - Research Site, Onesse-Laharie
  - Research Site, Oradour-sur-Vayres
  - Research Site, Orcines
  - Research Site, Orgères
  - Research Site, Orléans
  - Research Site, Orly
  - Research Site, Orry-la-Ville
  - Research Site, Orthez
  - Research Site, Oudon
  - Research Site, Oyonnax
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paillencourt
  - Research Site, Pantin
  - Research Site, Parcé-sur-Sarthe
  - Research Site, Parçay-Meslay
  - Research Site, Paris
  - Research Site, Parthenay
  - Research Site, Pau
  - Research Site, Peaugres
  - Research Site, Peltre
  - Research Site, Penmarch
  - Research Site, Percy
  - Research Site, Perpignan
  - Research Site, Perros-Guirec
  - Research Site, Pertuis
  - Research Site, Petite Ile
  - Research Site, Petite-Forêt
  - Research Site, Peyrat-le-Château
  - Research Site, Pélissanne
  - Research Site, Pénestin
  - Research Site, Pérenchies
  - Research Site, Pibrac
  - Research Site, Pignan
  - Research Site, Pisany
  - Research Site, Plabennec
  - Research Site, Plaisance-du-Touch
  - Research Site, Plan-de-Cuques
  - Research Site, Pleaux
  - Research Site, Plestin-les-Grèves
  - Research Site, Pleumeur-Gautier
  - Research Site, Ploeren
  - Research Site, Plombières-lès-Dijon
  - Research Site, Plouarzel
  - Research Site, Ploufragan
  - Research Site, Plourivo
  - Research Site, Plouvorn
  - Research Site, Plouzané
  - Research Site, Pocé-sur-Cisse
  - Research Site, Poissy
  - Research Site, Pont Ste Maxence
  - Research Site, Pont-de-Buis-lès-Quimerch
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pontailler-sur-Saône
  - Research Site, Pontault-Combault
  - Research Site, Pontcharra
  - Research Site, Pornic
  - Research Site, Port Leucate
  - Research Site, Port-de-Bouc
  - Research Site, Potigny
  - Research Site, Pradines
  - Research Site, Preignac
  - Research Site, Préchac
  - Research Site, Privas
  - Research Site, Prix-lès-Mézières
  - Research Site, Puget-Ville
  - Research Site, Pulnoy
  - Research Site, Puteaux
  - Research Site, Puttelange-aux-Lacs
  - Research Site, Quarouble
  - Research Site, Questembert
  - Research Site, Quiberon
  - Research Site, Quimper
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quincy-Voisins
  - Research Site, Rabastens-de-Bigorre
  - Research Site, Raismes
  - Research Site, Ramatuelle
  - Research Site, Ravières
  - Research Site, Rebais
  - Research Site, Reims
  - Research Site, Renazé
  - Research Site, Rezé
  - Research Site, Réding
  - Research Site, Ribemont
  - Research Site, Ribécourt-Dreslincourt
  - Research Site, Richemont
  - Research Site, Riedisheim
  - Research Site, Rieumes
  - Research Site, Rieupeyroux
  - Research Site, Riez
  - Research Site, Rilhac-Rancon
  - Research Site, Rillieux-la-Pape
  - Research Site, Rion-des-Landes
  - Research Site, Rixheim
  - Research Site, Robion
  - Research Site, Rochecorbon
  - Research Site, Rodez
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Rohrwiller
  - Research Site, Roisel
  - Research Site, Roissy-en-France
  - Research Site, Romainville
  - Research Site, Rombas
  - Research Site, Romorantin-Lanthenay
  - Research Site, Roncey
  - Research Site, Ronchin
  - Research Site, Rosières-en-Santerre
  - Research Site, Rosny-sous-Bois
  - Research Site, Rosny-sur-Seine
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Rouillac
  - Research Site, Royan
  - Research Site, Royaumeix
  - Research Site, Ruaux
  - Research Site, Rueil-Malmaison
  - Research Site, Ruelisheim
  - Research Site, Rully
  - Research Site, Ruy
  - Research Site, Sabres
  - Research Site, Sainpuits
  - Research Site, Sains-du-Nord
  - Research Site, Saint Georges Baillargeaux
  - Research Site, Saint Maximin La Ste Baume
  - Research Site, Saint-Affrique
  - Research Site, Saint-André-d'Apchon
  - Research Site, Saint-André-de-l'Eure
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-André-des-Eaux
  - Research Site, Saint-André-lez-Lille
  - Research Site, Saint-Arnoult-en-Yvelines
  - Research Site, Saint-Astier
  - Research Site, Saint-Aubin-des-Châteaux
  - Research Site, Saint-Aunès
  - Research Site, Saint-Avold
  - Research Site, Saint-Beauzire
  - Research Site, Saint-Benoît
  - Research Site, Saint-Bonnet-le-Château
  - Research Site, Saint-Chaffrey
  - Research Site, Saint-Claude-de-Diray
  - Research Site, Saint-Cyprien
  - Research Site, Saint-Denis
  - Research Site, Saint-Etienne
  - Research Site, Saint-Étienne-de-Baïgorry
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Étienne-du-Rouvray
  - Research Site, Saint-Étienne-les-Orgues
  - Research Site, Saint-Étienne-lès-Remiremont
  - Research Site, Saint-Fons
  - Research Site, Saint-Georges-du-Bois
  - Research Site, Saint-Germain-de-la-Coudre
  - Research Site, Saint-Girons
  - Research Site, Saint-Guénolé
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-du-Gard
  - Research Site, Saint-Jorioz
  - Research Site, Saint-Joseph
  - Research Site, Saint-Just-de-Claix
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Léger-en-Yvelines
  - Research Site, Saint-Louis
  - Research Site, Saint-Lô
  - Research Site, Saint-Martin-d'Hères
  - Research Site, Saint-Martin-d'Oney
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Martin-en-Haut
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-en-Gourgois
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Omer
  - Research Site, Saint-Paul-en-Chablais
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Philbert-de-Bouaine
  - Research Site, Saint-Pierre-d'Albigny
  - Research Site, Saint-Pierre-de-Chandieu
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-des-Fleurs
  - Research Site, Saint-Pierre-en-Val
  - Research Site, Saint-Pol-sur-Mer
  - Research Site, Saint-Porchaire
  - Research Site, Saint-Pourçain-sur-Sioule
  - Research Site, Saint-Priest
  - Research Site, Saint-Quentin
  - Research Site, Saint-Rambert-d'Albon
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Romain-de-Colbosc
  - Research Site, Saint-Sauveur-dAunis
  - Research Site, Saint-Savinien
  - Research Site, Saint-Savournin
  - Research Site, Saint-Sébastien-sur-Loire
  - Research Site, Saint-Sulpice-de-Royan
  - Research Site, Saint-Sylvain
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saint-Vallier
  - Research Site, Saint-Yorre
  - Research Site, Saintes
  - Research Site, Salbris
  - Research Site, Salernes
  - Research Site, Salies-du-Salat
  - Research Site, Salles
  - Research Site, Salles-Adour
  - Research Site, Salomé
  - Research Site, Sarre-Union
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sars-Poteries
  - Research Site, Saulnot
  - Research Site, Sault-lès-Rethel
  - Research Site, Savignac-les-Églises
  - Research Site, Savigneux
  - Research Site, Savigné-l'Évêque
  - Research Site, Savigny-sur-Orge
  - Research Site, Savonnières
  - Research Site, Schirmeck
  - Research Site, Scionzier
  - Research Site, Seclin
  - Research Site, Secondigny
  - Research Site, Sedan
  - Research Site, Seignosse
  - Research Site, Seloncourt
  - Research Site, Senones
  - Research Site, Seraincourt
  - Research Site, Sète
  - Research Site, Sèvres
  - Research Site, Sées
  - Research Site, Sérifontaine
  - Research Site, Sérignan
  - Research Site, Simiane-Collongue
  - Research Site, Six-Fours-les-Plages
  - Research Site, Sixt-sur-Aff
  - Research Site, Socx
  - Research Site, Soissons
  - Research Site, Soisy-sous-Montmorency
  - Research Site, Solliès-Pont
  - Research Site, Solre-le-Château
  - Research Site, Sorcy-Saint-Martin
  - Research Site, Soultz-sous-Forêts
  - Research Site, St-Malo
  - Research Site, Stains
  - Research Site, Ste Anne
  - Research Site, Ste Clotilde
  - Research Site, Ste Fereole
  - Research Site, Ste Fortunade
  - Research Site, Ste Foy de Peyrolieres
  - Research Site, Ste Foy La Grande
  - Research Site, Ste Livrade Sur Lot
  - Research Site, Ste Marie
  - Research Site, Ste Mere Eglise
  - Research Site, Ste Severe Sur Indre
  - Research Site, Ste Suzanne
  - Research Site, Strasbourg
  - Research Site, Sury-le-Comtal
  - Research Site, Talant
  - Research Site, Talence
  - Research Site, Tarascon
  - Research Site, Tarbes
  - Research Site, Tartas
  - Research Site, Téteghem
  - Research Site, Thérouanne
  - Research Site, Thiberville
  - Research Site, Thiel-sur-Acolin
  - Research Site, Thilouze
  - Research Site, Thionville
  - Research Site, Thuré
  - Research Site, Thurins
  - Research Site, Thyez
  - Research Site, Tiercé
  - Research Site, Til-Châtel
  - Research Site, Tincques
  - Research Site, Torcy
  - Research Site, Toufflers
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Touquin
  - Research Site, Tourcoing
  - Research Site, Tours
  - Research Site, Tourtour
  - Research Site, Traînel
  - Research Site, Traînou
  - Research Site, Trets
  - Research Site, Trégourez
  - Research Site, Tréguier
  - Research Site, Trignac
  - Research Site, Trith-Saint-Léger
  - Research Site, Troyes
  - Research Site, Tulle
  - Research Site, Turretot
  - Research Site, Uckange
  - Research Site, Uriménil
  - Research Site, Vabres-l'Abbaye
  - Research Site, Vailhauquès
  - Research Site, Valbonne
  - Research Site, Valence-d'Albigeois
  - Research Site, Valentigney
  - Research Site, Valff
  - Research Site, Vallauris
  - Research Site, Valras-Plage
  - Research Site, Vanault-les-Dames
  - Research Site, Vanves
  - Research Site, Varreddes
  - Research Site, Vasles
  - Research Site, Vaugneray
  - Research Site, Vauhallan
  - Research Site, Vaulx-en-Velin
  - Research Site, Vauvert
  - Research Site, Velleron
  - Research Site, Venarey-les-Laumes
  - Research Site, Vendeuil
  - Research Site, Vendôme
  - Research Site, Vennecy
  - Research Site, Verdelais
  - Research Site, Verdun
  - Research Site, Verfeil
  - Research Site, Verny
  - Research Site, Vers-Pont-du-Gard
  - Research Site, Versailles
  - Research Site, Vert-Saint-Denis
  - Research Site, Vélizy-Villacoublay
  - Research Site, Vénissieux
  - Research Site, Vieille-Église
  - Research Site, Vienne
  - Research Site, Vif
  - Research Site, Vigneux-sur-Seine
  - Research Site, Villard-Bonnot
  - Research Site, Villecresnes
  - Research Site, Villefagnan
  - Research Site, Villefranche-de-Lauragais
  - Research Site, Villefranche-de-Lonchat
  - Research Site, Villefranche-de-Rouergue
  - Research Site, Villejuif
  - Research Site, Villemeux-sur-Eure
  - Research Site, Villenave-d'Ornon
  - Research Site, Villeneuve-le-Roi
  - Research Site, Villeneuve-lès-Avignon
  - Research Site, Villeneuve-sur-Lot
  - Research Site, Villeneuve-Tolosane
  - Research Site, Villers-Bocage
  - Research Site, Villers-Bretonneux
  - Research Site, Villette-d'Anthon
  - Research Site, Villette-de-Vienne
  - Research Site, Villeurbanne
  - Research Site, Villeveyrac
  - Research Site, Villiers-sur-Marne
  - Research Site, Vinon-sur-Verdon
  - Research Site, Viry-Châtillon
  - Research Site, Vitré
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittefleur
  - Research Site, Voinémont
  - Research Site, Voiron
  - Research Site, Vouillé
  - Research Site, Voujeaucourt
  - Research Site, Vue
  - Research Site, Wambrechies
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Waziers
  - Research Site, Wignehies
  - Research Site, Yerville
  - Research Site, Yvré-le-Pôlin
  - Research Site, Zuydcoote